CLINICAL TRIAL: NCT03865186
Title: An Evaluation of a Psychoeducation Program for Emotion Identification and Expression in Individuals Diagnosed With Schizophrenia
Brief Title: An Evaluation of a Psychoeducation Program in Individuals Diagnosed With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Elif Aşık, principal investigator, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EAsik
Record Dates: First submitted 2019-02-26; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia
Keywords: Cognition; facial expression; facial recognition; psychiatric nursing; psychoeducation; schizophrenia
MeSH Terms: conditions — Schizophrenia; Facial Expression

STUDY DESIGN:
Intervention Model Description: This study was of quasi-experimental (pretest-posttest, with a control group) design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The program titled, "Psychoeducation Program for Emotion Identification and Expression in Those Diagnosed with Schizophrenia" was conducted with the patients in the intervention groups once a week for ten weeks.
  Interventions: Behavioral: Psychoeducation Program
- control group (Experimental): no intervention was applied to the control group
  Interventions: Behavioral: no intervention

INTERVENTIONS:
Behavioral: Psychoeducation Program — The program titled, "Psychoeducation Program for Emotion Identification and Expression in Those Diagnosed with Schizophrenia" was conducted with the patients in the intervention groups once a week for ten weeks.
  Arms: intervention group
Behavioral: no intervention
  Arms: control group

SUMMARY:
This study was conducted to explore the effect on social functionality of the psychoeducation program organized to guide individuals diagnosed with schizophrenia to identifying and recognize emotions in facial expressions. half of participants were assessed the psychoeducation program. other half of participants were used only measurement tests.

DETAILED DESCRIPTION:
The difficulties those diagnosed with schizophrenia have with facial identification and identifying emotions are closely associated with the adverse symptoms of the illness. Those diagnosed with schizophrenia need to be helped in forming interpersonal relations so that they can gain the skills needed to live in society.

ın this study the investigators prepared a psychoeducation program for individuals diagnosed with schizophrenia. The program titled, "Psychoeducation Program for Emotion Identification and Expression in Those Diagnosed with Schizophrenia" was conducted with the patients in the intervention groups once a week for ten weeks. On the other hand there were a control group which weren't be applied any intervention. The investigators applied some tests to intervention and control group three times ( before intervention, after intervention and three months after intervention). This study was conducted at three Community Mental Health Centers (CMHC's). The patients who met the study inclusion criterias were determined in these centers. Randomized psychoeducation and control groups were formed from these patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia according to DSM-IV
* over the age of 18

Exclusion Criteria:

* having cominication problems
* having another psychiatric disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Facial Emotion Identification | 15 minutes
  Facial Emotion Identification Test (FEIT) The test is in the form of a slide presentation of 19 black-and-white facial photographs displaying expressions of different emotions. Correct answers are rated 1, errors are scored 0. The highest possible score on the test is 19
Facial Emotion Discrimination | 20 minutes
  Facial Emotion Discrimination Test (FEDT) This consists of 30 pairs of black-and-white photographs depicting six main emotional states (happiness, sadness, anger, fear, surprise, embarrassment). The participant is asked to differentiate the photographs in each pair, determining whether the two facial expressions are the same or different. If the answer is correct, it is scored 1; if wrong, the score is 0. The highest possible score on the test is 30

SECONDARY OUTCOMES:
Personal and Social Performance | 20 minutes
  Personal and Social Performance Test (PSP) This is a 6-item Likert-type ranked assessment of four dimensions.The patient is first evaluated on the basis of the four dimensions and then the scores in these areas are entered into the score sheet on the basis of 10-point ranges from 10-100 according to the PSP assessment guidelines, assigning the patient a total PSP score. The higher scores indicate better functionality

CONTACTS AND LOCATIONS:
Overall Officials: Gül Ünsal, PhD, Study Director — Marmara University

IPD SHARING:
Plan to Share IPD: No
this study manuscript sended to an academic journal

REFERENCES:
- [Background] Allott KA, Rice S, Bartholomeusz CF, Klier C, Schlogelhofer M, Schafer MR, Amminger GP. Emotion recognition in unaffected first-degree relatives of individuals with first-episode schizophrenia. Schizophr Res. 2015 Feb;161(2-3):322-8. doi: 10.1016/j.schres.2014.12.010. Epub 2014 Dec 19. PMID 25533595
- [Background] Byrne LK, Pan L, McCABE M, Mellor D, Xu Y. Assessment of a six-week computer-based remediation program for social cognition in chronic schizophrenia. Shanghai Arch Psychiatry. 2015 Oct;27(5):296-306. doi: 10.11919/j.issn.1002-0829.215095. PMID 26977127
- [Background] Calvo A, Moreno M, Ruiz-Sancho A, Rapado-Castro M, Moreno C, Sanchez-Gutierrez T, Arango C, Mayoral M. Psychoeducational Group Intervention for Adolescents With Psychosis and Their Families: A Two-Year Follow-Up. J Am Acad Child Adolesc Psychiatry. 2015 Dec;54(12):984-90. doi: 10.1016/j.jaac.2015.09.018. Epub 2015 Oct 13. PMID 26598473
- [Background] Cohen AS, Minor KS. Emotional experience in patients with schizophrenia revisited: meta-analysis of laboratory studies. Schizophr Bull. 2010 Jan;36(1):143-50. doi: 10.1093/schbul/sbn061. Epub 2008 Jun 17. PMID 18562345
- [Background] Combs DR, Chapman D, Waguspack J, Basso MR, Penn DL. Attention shaping as a means to improve emotion perception deficits in outpatients with schizophrenia and impaired controls. Schizophr Res. 2011 Apr;127(1-3):151-6. doi: 10.1016/j.schres.2010.05.011. Epub 2010 Jun 8. PMID 20570490
- [Background] Combs DR, Tosheva A, Penn DL, Basso MR, Wanner JL, Laib K. Attentional-shaping as a means to improve emotion perception deficits in schizophrenia. Schizophr Res. 2008 Oct;105(1-3):68-77. doi: 10.1016/j.schres.2008.05.018. Epub 2008 Jun 27. PMID 18585899
- [Background] Drusch K, Stroth S, Kamp D, Frommann N, Wolwer W. Effects of Training of Affect Recognition on the recognition and visual exploration of emotional faces in schizophrenia. Schizophr Res. 2014 Nov;159(2-3):485-90. doi: 10.1016/j.schres.2014.09.003. Epub 2014 Sep 20. PMID 25248938
- [Background] Gaudelus B, Virgile J, Geliot S; GAIA/RECOS Study Team; Franck N. Improving Facial Emotion Recognition in Schizophrenia: a Controlled Study Comparing Specific and Attentional Focused Cognitive Remediation. Front Psychiatry. 2016 Jun 21;7:105. doi: 10.3389/fpsyt.2016.00105. eCollection 2016. PMID 27445866
- [Background] Gur RC, Gur RE. Social cognition as an RDoC domain. Am J Med Genet B Neuropsychiatr Genet. 2016 Jan;171B(1):132-41. doi: 10.1002/ajmg.b.32394. Epub 2015 Nov 26. PMID 26607670
- [Background] Hooker CI, Bruce L, Fisher M, Verosky SC, Miyakawa A, Vinogradov S. Neural activity during emotion recognition after combined cognitive plus social cognitive training in schizophrenia. Schizophr Res. 2012 Aug;139(1-3):53-9. doi: 10.1016/j.schres.2012.05.009. Epub 2012 Jun 12. PMID 22695257
- [Background] Huang CL, Hsiao S. The Functional Significance of Affect Recognition, Neurocognition, and Clinical Symptoms in Schizophrenia. PLoS One. 2017 Jan 18;12(1):e0170114. doi: 10.1371/journal.pone.0170114. eCollection 2017. PMID 28099444
- [Background] Kerr SL, Neale JM. Emotion perception in schizophrenia: specific deficit or further evidence of generalized poor performance? J Abnorm Psychol. 1993 May;102(2):312-8. doi: 10.1037//0021-843x.102.2.312. PMID 8315144
- [Background] Kring AM, Elis O. Emotion deficits in people with schizophrenia. Annu Rev Clin Psychol. 2013;9:409-33. doi: 10.1146/annurev-clinpsy-050212-185538. Epub 2012 Dec 10. PMID 23245340
- [Background] Lindenmayer JP, McGurk SR, Khan A, Kaushik S, Thanju A, Hoffman L, Valdez G, Wance D, Herrmann E. Improving social cognition in schizophrenia: a pilot intervention combining computerized social cognition training with cognitive remediation. Schizophr Bull. 2013 May;39(3):507-17. doi: 10.1093/schbul/sbs120. Epub 2012 Nov 3. PMID 23125396
- [Background] Marsh PJ, Luckett G, Russell T, Coltheart M, Green MJ. Effects of facial emotion recognition remediation on visual scanning of novel face stimuli. Schizophr Res. 2012 Nov;141(2-3):234-40. doi: 10.1016/j.schres.2012.08.006. Epub 2012 Sep 5. PMID 22959743
- [Background] Morosini PL, Magliano L, Brambilla L, Ugolini S, Pioli R. Development, reliability and acceptability of a new version of the DSM-IV Social and Occupational Functioning Assessment Scale (SOFAS) to assess routine social functioning. Acta Psychiatr Scand. 2000 Apr;101(4):323-9. PMID 10782554
- [Background] Rose A, Vinogradov S, Fisher M, Green MF, Ventura J, Hooker C, Merzenich M, Nahum M. Randomized controlled trial of computer-based treatment of social cognition in schizophrenia: the TRuSST trial protocol. BMC Psychiatry. 2015 Jul 3;15:142. doi: 10.1186/s12888-015-0510-1. PMID 26138715